CLINICAL TRIAL: NCT02366572
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 1 - Acute Effects of Pulse Ingredients in Snack Products on Appetite, Blood Glucose, and Food Intake in Adults - Study 2
Brief Title: PERFECT Project - Part 1 - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:114-3
Record Dates: First submitted 2014-12-17; First posted 2015-02-19 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention
MeSH Terms: interventions — Pea Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cereal control (Placebo Comparator): 100% Wheat Flour
  Interventions: Other: Control
- Cereal with pea protein (Experimental): Pea protein
  Interventions: Other: Pea protein
- Cereal with pea starch (Experimental): Pea starch
  Interventions: Other: Pea starch
- Cereal w/ pea starch + pea fibre: 5g (Experimental): Pea starch + pea fibre: 5g
  Interventions: Other: Pea fibre + pea starch
- Cereal w/ pea protein + pea starch: 10g (Experimental): Pea protein + pea starch: 10g
  Interventions: Other: Pea protein + pea starch
- Cereal w/ pea protein + pea fibre + pea starch: 20g (Experimental): Pea protein + pea fibre + pea starch: 20g
  Interventions: Other: Pea fibre + pea starch + pea protein

INTERVENTIONS:
Other: Control — Non pulse extruded cereal
  Arms: Cereal control
Other: Pea protein — Pulse extruded cereal
  Arms: Cereal with pea protein
Other: Pea starch — Pulse extruded cereal
  Arms: Cereal with pea starch
Other: Pea fibre + pea starch — Pulse extruded cereal
  Arms: Cereal w/ pea starch + pea fibre: 5g
Other: Pea protein + pea starch — Pulse extruded cereal
  Arms: Cereal w/ pea protein + pea starch: 10g
Other: Pea fibre + pea starch + pea protein — Pulse extruded cereal
  Arms: Cereal w/ pea protein + pea fibre + pea starch: 20g

SUMMARY:
The objectives are to test the acute effects of different cereals containing pulse ingredients on: 1) post-prandial blood glucose, insulin and appetite for two hours, and 2) food intake two hours following consumption of pulse products.

We hypothesize that cereals containing pulse ingredients will lead to lower blood glucose, insulin, appetite and food intake responses compared to non-pulse cereals.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Competitive sports or athletic training at a high intensity
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.
* Those unable to walk for an hour continuously

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0 - 200 min
  Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits
Food Intake | at 120 min
  Measured by VAS questionnaire
Subjective Appetite | 0-200 min
  Motivation-to-eat VAS questionnaire

SECONDARY OUTCOMES:
Palatability of treaments and meal | 5 and 140 minutes
  Measured by VAS questionnaire
Physical comfort | 0 - 200 min
  Measured by VAS questionnaire
Energy/fatigue | 0-200 min
  Measured by VAS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals

REFERENCES:
- [Derived] Johnston AJ, Mollard RC, Dandeneau D, MacKay DS, Ames N, Curran J, Bouchard DR, Jones PJ. Acute effects of extruded pea fractions on glycemic response, insulin, appetite, and food intake in healthy young adults, results of a double-blind, randomized crossover trial. Appl Physiol Nutr Metab. 2021 Sep;46(9):1126-1132. doi: 10.1139/apnm-2020-0571. Epub 2021 Mar 4. PMID 33661714